CLINICAL TRIAL: NCT01406730
Title: Effect of 16 Weeks of Running Exercise on Parameters Related to the Cardiovascular System, Blood and Muscle in Untrained Males 30-50 Years Old. A Randomized Controlled Study
Brief Title: Running Effect on Cardiovascular and Muscular Parameters
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: University of Erlangen-Nürnberg (Other); Institute of Physical Education and Sports Sciences (Other); Klinikum Nürnberg (Other)
Responsible Party: Principal Investigator, Wolfgang Kemmler, Prof. Dr., University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FAU-IMP-4463
Record Dates: First submitted 2011-07-18; First posted 2011-08-01 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Males; Untrained; 30-50 Years Old; Healthy
Keywords: running exercise; cardiac hypertrophy; blood; maximum oxygen uptake; intervention; untrained; males
MeSH Terms: conditions — Cardiomegaly | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- exercise (Experimental): 16 weeks of running exercise
  Interventions: Other: exercise
- control (No Intervention)

INTERVENTIONS:
Other: exercise — 16 week of periodized progressive running exercise 2-4 times/week
  Arms: exercise

SUMMARY:
The purpose of the study is to determine the effect of 16 weeks of running exercise on various parameters related to heart, vascular systems, blood, and muscle in untrained males 30-50 years old.

Further, the investigators assess which of the above mentioned parameters may explain the increase of running performance most accurate.

ELIGIBILITY:
Inclusion Criteria:

* males
* untrained (< 2 endurance exercise sessions/week)
* 30-50 years old

Exclusion Criteria:

* pathological changes of the heart
* inflammable diseases
* medication/diseases affecting cardiovascular system and muscle
* very low physical capacity (< 100 Watt at ergometry)
* obesity (BMI > 30 kg/m2)
* more than 2 weeks of absence during the interventional period
* more than 2 exercise session beside the intervention
* contraindication related to MRI-assessment (i.e. claustrophobia, magnetizable intracorporal artefacts)

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
myocardial mass/stroke volume | 4 month
  Atrial and ventricular volume and mass indexes were assessed by magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
maximal oxygen uptake | 4 month
  maximal oxygen uptake during running
Resting metabolic rate | 4 month
  Adaptation of resting metabolic rate to running exercise
muscle strength/power | 4 month
  Isometric muscle strength of the leg extensors Leg power as assessed by counter movement jump
myocardial volume | 4 month
  Functional and morphologic parameters of the heart as assessed by echocardiography
Intima media thickness | 4 month
  Carotid intima media thickness by high-resolution ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lell, MD, Study Director — Departement of Radiology, Division of Cardiology, University of Erlangen-Nurnberg; Michael Scharf, MD, Principal Investigator — Departement of Radiology, Division of Cardiology; Willi A Kalender, PhD, Study Chair — Institute of Medical Physics, University of Erlangen, Germany; Michael Uder, MD, Study Chair — Departement of Radiology, University of Erlangen-Nurnberg; Wolfgang Kemmler, PhD, Study Director — Institute of Medical Physics, University of Erlangen-Nurnberg, Germany; Simon von Stengel, PhD, Principal Investigator — University of Erlangen-Nürnberg Medical School
Locations (3):
- Germany (3):
  - Institute of Medical Physics, University of Erlangen-Nurnberg, Erlangen
  - Institute of Physical Education and Sport Sciences, Erlangen
  - Departement of Radiology, University of Erlangen-Nurnberg, Erlangen

REFERENCES:
- [Background] Scharf M, Brem MH, Wilhelm M, Schoepf UJ, Uder M, Lell MM. Atrial and ventricular functional and structural adaptations of the heart in elite triathletes assessed with cardiac MR imaging. Radiology. 2010 Oct;257(1):71-9. doi: 10.1148/radiol.10092377. Epub 2010 Aug 31. PMID 20807850
- [Derived] Tuttor M, von Stengel S, Kohl M, Lell M, Scharf M, Uder M, Wittke A, Kemmler W. High Intensity Resistance Exercise Training vs. High Intensity (Endurance) Interval Training to Fight Cardiometabolic Risk Factors in Overweight Men 30-50 Years Old. Front Sports Act Living. 2020 Jun 16;2:68. doi: 10.3389/fspor.2020.00068. eCollection 2020. PMID 33345059
- [Derived] Scharf M, Schmid A, Kemmler W, von Stengel S, May MS, Wuest W, Achenbach S, Uder M, Lell MM. Myocardial adaptation to high-intensity (interval) training in previously untrained men with a longitudinal cardiovascular magnetic resonance imaging study (Running Study and Heart Trial). Circ Cardiovasc Imaging. 2015 Apr;8(4):e002566. doi: 10.1161/CIRCIMAGING.114.002566. PMID 25873721
- See also: homepage of the Institute of Medical Physical with study informations. — http://www.imp.uni-erlangen.de/